CLINICAL TRIAL: NCT00563602
Title: Randomized and Controlled Study of Endoscopic Ligation, Nadolol and Isosorbide Mononitrate vs Endoscopic Ligation and Nadolol Alone, or Associated With Isosorbide Mononitrate or Prazosin, Depending of the Hemodinamyc Response
Brief Title: Treatment for Prevention of Variceal Rebleeding Guided by the Hemodynamic Response
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CONHEMO-2006; EudraCT 2007-002237-37
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Portal Hypertension; Complications of Cirrhosis
Keywords: Portal hypertension; Prevention of rebleeding; Complications of cirrhosis; Portal hemodynamic; Prazosine; Nadolol; isosorbide mononitrate
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Standard Therapy: Endoscopic ligation (LEV) + Nadolol + Isosorbide mononitrate (MNI)(drugs carefully titrated until achieve maximum tolerated dose)
  Interventions: Other: Hemodynamic guided therapy
- 1 (Experimental): Hemodynamic guided therapy:
  1) LEV + Nadolol. HVPG measurement: if response, no changes, if not, switch to 2) LEV + Nadolol + MNI. HVPG measurement: if response, no changes, if not, switch to: 3) LEV + Nadolol + Prazosin. (drugs carefully titrated until achieve maximum tolerated dose)
  Interventions: Other: Hemodynamic guided therapy

INTERVENTIONS:
Other: Hemodynamic guided therapy — To switch two or more different treatments for the prevention of variceal rebleeding according to the hemodynamic response. All patients in the experimental group will begin by:
  1) LEV + Nadolol. HVPG measurement: if response, no changes, if not, switch to 2) LEV + Nadolol + MNI. HVPG measurement: if response, no changes, if not, switch to: 3) LEV + Nadolol + Prazosin. (drugs carefully titrated until achieve maximum tolerated dose)

SUMMARY:
This is a prospective trial of random distribution, open, parallel group, in which patients with esophagic variceal bleeding will be randomized into two treatment groups, after controlling acute bleeding. All patients received standard medical therapy with b-blockers and endoscopic ligation (LEV) of esophageal varices.

The control group will be assigned to receive LEV + Nadolol + MNI. The experimental group will be assigned to receive treatment according to the hemodynamic response.

All patients included in the experimental group received LEV and pharmacological treatment nadolol alone or combined with MNI or Prazosin (PZ)

DETAILED DESCRIPTION:
This is a prospective trial of random distribution, open, parallel group, in which patients with esophagic variceal bleeding will be randomized into two treatment groups, after controlling acute bleeding. All patients received standard medical therapy with b-blockers and endoscopic ligation (LEV) of esophageal varices.

The control group will be assigned to receive LEV + Nadolol (N) + Isosorbide Mononitrate (MNI) The experimental group will be assigned to receive treatment according to the hemodynamic response.

All patients included in the experimental group received LEV and pharmacological treatment nadolol alone or combined with MNI or Prazosin (PZ)

A hepatic hemodynamic study will be performed to patients in both groups, at baseline (In which basal values and acute b-blockers response will be assessed), and a second study at the 3 rd -4 th week after the drug therapy start, after the titration of the doses.

In the experimental group, responders to the acute administration of b-blockers will receive LEV + Nadolol alone, and those patients with no response will receive LEV + N + MNI, and another hemodynamic study will be performed 3 rd -4 th week after the drug therapy start, after the titration of the doses, to assess response. The non-responders in this control study will switched to LEV+ N + PZ, and a 3erd hemodynamic study will be performed.

Randomization will be stratified according to the degree of hepatic insufficiency, assessed by the Child-Pugh classification (classes A and B vs C)

ELIGIBILITY:
Inclusion Criteria:

* All the patients admitted in emergencies in which 1) with gastrointestinal bleeding due to esophageal varices assessed by endoscopy, will be included.
* We define esophagic variceal bleeding as the endoscopic finding of any the following signs: 1) active variceal bleeding 2) clot or platelet cluster or 3 ) esophageal varices associated to red blood in esophagogastric lumen in the absence of other sources of bleeding.
* Clinical criteria and / or analytical, ultrasound and / or liver biopsy consistent with the diagnosis of liver cirrhosis.
* Written informed consent to participate in the study.
* Patients in fertile age should use barrier methods to prevent pregnancy during the entire study. The pregnancy test prior to the study must be negative

Exclusion Criteria:

* Age <18 or> 80 years.
* Patients not eligible for active treatment due to any underlying morbid condition (terminals). Here are included those patients with advanced liver disfunction (Child-Pugh >) or any patient with life expectancy < 6 mo.
* Refuse to participate in the study.
* Bleeding due to causes other than the esophageal varices.
* Prior inclusion in this study.
* Failure in the control of the acute bleeding (index episode).
* Pretreatment through elective LEV program, sclerotherapy or combined β- blockers plus nitrates, or portosystemic shunt (surgical or percutaneous).
* Contraindication for β- blockers and MNI (not exclude patients with contraindication for one of these drugs) or endoscopic procedures.
* Pregnancy.
* Presence multiple hepatocellular carcinoma or only diameter > 5 cm.
* Portal vein thrombosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-08; Study Completion 2007-11 (Estimated)

PRIMARY OUTCOMES:
Rebleeding | 1-2 Years

SECONDARY OUTCOMES:
Survival | 1-2 Years
Adverse effects | 1-2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Candid Villanueva, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- HospitalSCSP, Barcelona, Barcelona, Spain